CLINICAL TRIAL: NCT00791986
Title: Effects of Loaded Breathing Training on Blood Pressure in Essential Hypertensive Patients
Brief Title: Loaded Breathing Training in Essential Hypertension
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of study time and budget permission
Sponsor: Khon Kaen University (Other)
Collaborators: Thai health promotion foundation. (Unknown)
Responsible Party: Principal Investigator, Benjarat Sangthong, Faculty of associated medical science, Khon Kaen University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: KKU-475090015-0
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Essential Hypertension
Keywords: Breathing exercise; blood pressure; hypertension
MeSH Terms: conditions — Essential Hypertension; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control (No Intervention): The patients in this control group do not conduct any breathing training.
- ULB (Experimental): The patients conduct controlled slow breathing training using the WPTB device without inspiratory resistance.
  Interventions: Device: ULB , LB
- LB (Experimental): The patients breath in against resistance using WPTB device.
  Interventions: Device: ULB , LB

INTERVENTIONS:
Device: ULB , LB — ULB: The patients breath in slowly without resistance via the water pressure threshold breathing (WPTB) device, 30 min/day, 7 days/week for 8 weeks.
  LB : The patients breath in slowly against resistance of 20 cmH2O provided by the water pressure threshold breathing (WPTB) device, 30 min/day, 7 days/week for 8 weeks.
  Other Names: Guided breathing training; Paced breathing training; Controlled breathing training
  Arms: LB; ULB

SUMMARY:
The purpose of this study is to determine whether adding load to slow controlled breathing training could enhance blood pressure lowering in patients with essential hypertension.

DETAILED DESCRIPTION:
Hypertension (HT) is one of the major risk of cardiovascular diseases and cost of pharmacological treatment is a very high. Lifestyle modification is the first trial in stage 1 hypertension before commencing pharmacological treatment and a co-treatment with drug in hypertensive patient. Slow paced breathing training and physical training has been shown to reduce both systolic and diastolic blood pressure in HT. Moreover loaded breathing was reported to be able to decrease blood pressure in healthy. Loaded slow breathing training may enhance the antihypertensive effect of slow paced breathing.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of essential hypertension stage I-II

Exclusion Criteria:

* Respiratory disease
* Diabetes mellitus
* Heart disease
* Renal disease
* Cerebrovascular disease
* Dyslipidemia
* Pregnancy

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-05; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Home blood pressure | Pre- and post - 8 weeks of intervention at rest

SECONDARY OUTCOMES:
Office blood pressure | Pre- and post- 8 weeks of intervention at rest
Exercising blood pressure | Blood pressure during exercise at pre- and post-8 weeks of intervention
Heart rate variability | Heart rate variability at pre-and post- 8 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Chulee U Jones, Ph.D., Study Chair — Department of Physical Therapy, Faculty of Associated Medical Sciences, Khon Kaen University.; Benjarat Sangthong, M.Sc., Principal Investigator — Faculty of Physical Therapy, Rungsit University
Locations (1):
- Cardiopulmonary Physical Therapy Research Room, Faculty of Asociated Medical Sciences, Khon Kaen University., Khon Kaen, Thailand

REFERENCES:
- [Background] - Seals DR, Suwarno NO, Joyner MJ et al.Respiratory modulation of muscle sympathetic nerve activity in intact and lung denervated humans. Circulation Research 72(2): 440-454,1993. - Rosenthal T, Alter A, Peleg E, Gavish B. Device-guided breathing exercises reduce blood pressure: ambulatory and home measurements. Am J Hypertens 14(1):74-76,2001. - Viskoper R, Shapira I, Priluck R et al.Nonpharmacologic treatment of resistant hypertensive by device-guided slow breathing exercises. Am J Hypertens 16(6): 484-487,2003. - Grossman E, Grossman A, Schein MH et al.Breathing-control lowers blood pressure. J Hum Hypertens 15(4): 263-269,2001. - Viskoper R, Shapira I, Priluck R et al.Nonpharmacologic treatment of resistant hypertensive by device-guided slow breathing exercises. Am J Hypertens 16(6):484-487,2003 - Meles E, Giannattasio C, Failla M. et al.Non-pharmacologic treatment of hypertension by respiratory exercise in the home setting. Am J Hypertens 17(4):370-374,2004.